CLINICAL TRIAL: NCT02648360
Title: Evaluation of a Text Messaging Program for Physical Activity and Healthy Eating for Underserved Hispanic Patients
Brief Title: Text Messaging for Physical Activity & Healthy Eating
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Mark Stoutenberg, Research Assistant Professor, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 20151048
Record Dates: First submitted 2016-01-05; First posted 2016-01-07 (Estimated); Last update posted 2016-12-28 (Estimated); Status verified 2016-12

CONDITIONS: Overweight
Keywords: exercise; diet; patients, underserved; text messaging
MeSH Terms: conditions — Overweight; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Text Messaging Intervention Arm (Experimental): Participants will be enrolled in either a dietary or physical activity text messaging program. The dietary program will include nutritional education, reading nutrition labels, portion control, making lifestyle changes, finding social support, and identifying triggers. The physical activity program will provide information on the benefits of physical activity, exercise tips, and encouragement to live more active lifestyles. The programs have limited interactive capability; patients will be asked to respond to specific questions, but questions asked by the participants will be answered with an automated message asking them to contact their health care provider.
  Interventions: Behavioral: Text Messaging

INTERVENTIONS:
Behavioral: Text Messaging — The content of the program will be delivered via 3 weekly text messages over a 4 month period of time.

SUMMARY:
Hispanics share a disproportionate burden of several of the nation's leading chronic diseases caused by poor lifestyle habits such as sedentary behavior and poor quality nutrition intake. This project will design, implement and evaluate the delivery and effectiveness of an existing health promotion text messaging program focused on increasing physical activity and improving dietary behaviors among medically underserved Hispanic patients. Adult Hispanic patients referred by their healthcare provider at a local free community health clinic will be invited to participate in the 4-month long study. Patients who agree to participate will be sent health promotion text messages and will complete a brief pre-post assessment battery. Patients who do not send an initial enrollment text (to agree to participate) will receive a follow up telephone call from the research team to encourage participation. Evaluations will consist of: (1) physician referral rates; (2) patient enrollment rates; (3) demographic differences (gender, age) in participants/non-participants; and (4) pre-post changes in levels of physical activity and quality dietary intake will be conducted. The results of this study will provide a better understanding of the feasibility and effectiveness of implementing referral-based text messaging programs among medically underserved Hispanic patients at high risk for chronic diseases.

DETAILED DESCRIPTION:
Referral Process When a patient at the participating free community health clinic sees their health care provider, they will be given a referral card with information on how to enroll in the text messaging program. The referral will also be recorded in the patient's electronic health record. Health care providers will be encouraged to recommend the program to all their patients who they feel will benefit from improving their activity levels or dietary habits. Patients who receive referral cards (i.e., clearance) for either text messaging program will have the choice of programs to enroll in. If a healthcare provider feels that a patient is not capable of participating in one of the text messaging interventions (i.e., due to a dietary restriction or physical limitation) they will be given only the referral card to which they are cleared to participate. Patients will be asked to text the number on the referral card if they are interested in participating in the text messaging program (passive recruitment process). Patients who text the number on the referral card will receive an automated reply indicating that they will be contacted within 1-2 days. A research team member will call the patient back to explain the text messaging program and initiate the enrollment process.

Patients who do not initially enroll by texting the number on the card will receive a follow up call by a clinic employee or volunteer approximately one to two weeks after the health care provider provides that patient with a referral (active recruitment process). The call will re-introduce the patient to the text messaging program and encourage their participation. If the patient agrees to enroll, they will be referred to the research team to initiate the enrollment process.

Data on the referral process (number of patients referred, referring physicians, etc.) may be shared with the research team at the discretion of the health clinic leadership. Shared information will be de-identified so that the research team will not be able to identify patients of the clinic.

Enrollment Process Patients that agree to participate in the program will be contacted by the research team. The patients will then be provided with an introduction to the study, the risks and benefits of participating, and asked to provide their verbal consent (see the "Verbal Consent" document in the Consent section of the protocol) agreeing to participate in the study. Following their verbal consent, eligible participants will be asked a number of questions about their demographic information, physical activity levels, and dietary habits (see the "Participant Questionnaire" document upload in the Supporting Document section).

At this point, the research team member will enroll the patient in the text messaging intervention. Participants will have the option of enrolling in the Physical Activity program (which focuses primarily on physical activity, but does include some dietary information) or the Nutrition program (which focuses primarily on nutrition, but does include some physical activity information) depending on the referral that they received as described above. Patients will be enrolled to the text messaging program on a rolling process throughout the study period.

If, during the enrollment process a patient declines to participate, they will be asked for their feedback on participating in the study (see the "Non-Participation Questions" document uploaded in the Supporting Document section) to seek information to improve the program and recruitment of participants in the future.

Text Messaging Program The text messaging programs to be used in this study were developed by Care Message, a non-profit organization based in San Francisco, CA. Care Message offers a cloud-based platform with options for several text messaging programs in English or Spanish on various topics such as health behavior change, chronic disease management, women's care, and preventive care. Programs last from 1 to 12 months, and consist of three weekly automated, culturally adapted, and interactive text messages designed to increase knowledge, self-efficacy, and improve health behaviors.

Study Assessments Evaluation of the effectiveness of the text messaging program will be conducted at baseline and at the completion of the 4-month intervention. An identical assessment protocol will be conducted at both time points to assess changes in eating habits and activity levels. Additionally, a participant satisfaction questionnaire will be conducted with study completers at the end of the intervention

ELIGIBILITY:
Inclusion Criteria:

* Spanish speaking adults
* Have a cell phone that they are able to use to send and receive text messages
* Basic level of literacy (i.e., ability to read text messages)
* Patients at the free community health clinic, who had an appointment with a physician during the study recruitment period
* Clearance by physician to participate (i.e., provision of referral card by physician is equivalent to medical clearance)

Exclusion Criteria:

* Pregnant women, children, or any other individuals that the physician deems not suitable for participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-01; Primary Completion 2016-05 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Mean change in activity levels as assessed by the Godin Leisure-Time Exercise Questionnaire | Change in physical activity levels from baseline at 4 months
  The Godin Leisure-Time Exercise Questionnaire has been found to be appropriate for assessing leisure time activity in a community setting with two week test-retest reliability coefficients of 0.48 for mild, 0.46 for moderate, and 0.94 for strenuous exercise. The questionnaire is brief, easily administered, reliable, and demonstrates concurrent validity with other tools.
Mean change in dietary habits as assessed by the Starting the Conversation Scale | Change in dietary habits from baseline at 4 months
  Starting The Conversation (STC) is a simplified screening instrument designed for non-dietitians in clinical practices for assessment and counseling. It identifies dietary patterns and was derived from a validated 54-item instrument.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Stoutenberg, PhD, MSPH, Principal Investigator — University of Miami

IPD SHARING:
Plan to Share IPD: No